CLINICAL TRIAL: NCT01158014
Title: Fibrin Glue vs. Vicryl Suture in Pterygium Surgery With Conjunctival Auto-graft
Brief Title: Fibrin Glue vs. Suture in Pterygium Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Guy Ben-Simon, MD (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Guy Ben-Simon, MD, Prof, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-5033-GB-CTIL
Record Dates: First submitted 2010-07-04; First posted 2010-07-08 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Conjunctival Autograft
Keywords: pterygium; conjunctival graft; recurrence; primary pterygium
MeSH Terms: conditions — Pterygium; Recurrence | interventions — Fibrin Tissue Adhesive; Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Glue, surgery (Experimental): Conjunctival autograft will be glued using fibrin glue to pterygia bed after removal
  Interventions: Procedure: Fibrin Glue, Quixil
- Control (Active Comparator): Conjunctival autograft will be sutured using 10/0 vicryl sutures to pterygia bed after removal
  Interventions: Procedure: Suture

INTERVENTIONS:
Procedure: Fibrin Glue, Quixil — quixil 0.1 ml
  Arms: Fibrin Glue, surgery
Procedure: Suture — vicryl 10/0
  Arms: Control

SUMMARY:
The use of Fibrin glue to place conjunctival graft will be as effective as suturing the graft, but will require much less operative time and will be better tolerated by the patients.

DETAILED DESCRIPTION:
Pterygium surgery requires removal of the pterygia from cornea and conjunctiva and an additional technique to prevent recurrence which may be as high as 50%.

Suturing a conjunctival auto-graft has become one of the most popular and effective methods in preventing recurrence. However suturing requires long operative time (10-20 minutes with removal alone less than 5 minutes) and requires sutures removal after 1-2 weeks which is very inconvenient to the patient.

Using Fibrin Glue (Quixil) has been used in several places in pterygium surgery and we believe it will be as effective as suturing the graft, will use much less OR time (reduce surgery time from 40 minutes to 20-25 minutes) and will be less expensive since 2 ml glue (around 80US$) suffice for 10 cases, while one vicryl suture costs around 34 US$.

ELIGIBILITY:
Inclusion Criteria:

* primary pterygium
* healthy subject
* ability to attend follow-up visits

Exclusion Criteria:

* recurrent pterygium
* underwent previous surgery / intervention to treat pterygium
* ocular surface disease 0 minor

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pterygium recurrence | one year
  Recurrence normally occurs 1-6 months after surgery. Success is achieved if ptergium does not recur after one year.

SECONDARY OUTCOMES:
operation time | one year
  suturing a conjunctival graft takes 15-10 minutes while gluing only 5 minutes, we believe that by lowering OR time, total costs of surgery are less

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

REFERENCES:
- [Result] Ratnalingam V, Eu AL, Ng GL, Taharin R, John E. Fibrin adhesive is better than sutures in pterygium surgery. Cornea. 2010 May;29(5):485-9. doi: 10.1097/ICO.0b013e3181c29696. PMID 20308876
- [Result] Por YM, Tan DT. Assessment of fibrin glue in pterygium surgery. Cornea. 2010 Jan;29(1):1-4. doi: 10.1097/ICO.0b013e3181a38fda. PMID 19907303
- [Result] Hall RC, Logan AJ, Wells AP. Comparison of fibrin glue with sutures for pterygium excision surgery with conjunctival autografts. Clin Exp Ophthalmol. 2009 Aug;37(6):584-9. doi: 10.1111/j.1442-9071.2009.02105.x. PMID 19702708